CLINICAL TRIAL: NCT06984211
Title: Cardio Alpha - Vibrometer Based Pulse Wave Analysis for Arterial Stiffness and Ischemic Heart Disease Risk Assessment
Brief Title: Vibrometer Based Pulse Wave Analysis for Arterial Stiffness and Ischemic Heart Disease Risk Assessment
Status: Recruiting | Type: Observational
Sponsor: HJN Sverige AB/Neko Health (Industry)
Responsible Party: Sponsor
Other Study IDs: CRD-P3-LMV_CIP-220623
Record Dates: First submitted 2023-08-01; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Hypertension; Ischemic Heart Disease; Valvular Heart Disease; Heart Failure; Diabetes
MeSH Terms: conditions — Hypertension; Myocardial Ischemia; Heart Valve Diseases; Heart Failure; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patient_cohort: Adult patients mainly from a primary care cohort. All patients visiting the clinical sites, seeking care, or as separately invited, are offered to participate in this investigation. This includes sub-groups of patients with hypertension, valvular disease or risk for IHD. All participants undergo at least one examination with the investigational device (Cardio P3) at initial visit.

SUMMARY:
This clinical investigation will evaluate a novel contactless technology for assessing arterial stiffness and explore its potential in assessment of risk for and development of cardiovascular disease.

The main aims of the study are:

1. To assess device and method performance for assessment of arterial stiffness and cardiovascular risk, on a prospective primary care cohort.
2. To see if precision may be added in CVD risk assessment through a multi-modal approach, combining data on macro- and micro-circulatory function.

DETAILED DESCRIPTION:
Arterial stiffness, commonly assessed as pulse wave velocity (PWV), is a marker of aging of the cardio-vascular system strongly associated with hypertension and increased risk for and development of cardiovascular disease.

This clinical investigation aims at evaluating the clinical safety, performance and potential value of a novel laser-radar-based vibrometer technology, for the assessment of arterial stiffness and to explore correlations of various measurements made with the technology with risk and development of cardiovascular disease, specifically ischemic heart disease, hypertension and aortic valve pathology.

The study participants mainly consist of a prospective primary care population, that undergo an investigation (including vibrometer and microwave radar assessment, blood pressure, ECG and ankle-brachial index) at a primary care visit. An extended investigation (including vibrometer assessment, cardiovascular ultrasound and other reference methods for pulse wave velocity and cardiovascular risk assessment) will be offered to participants judged to have an increased risk of cardiovascular disease in the primary care population, or for separately invited subjects with increased cardiovascular risk, known valvular disease, or as healthy controls. Repeated yearly measurements plan to be performed in interested subjects.

A subset of the participants will undergo a contactless multi-modal investigation which includes combining data from the current study with contactless spatial frequency domain data from the investigation "Spectrum 1" (CIV ID: CIV-22-07-039907). The hypothesis is that CVD risk assessment may be improved through a multi-modal approach, combining data on both macro- and micro-circulatory function.

A subset of the data will be used to evaluate the association between the prevalence of hypertension and total peripheral resistance, as well as cardiac output.

The study is of exploratory character with many analyses; however, the main outcomes are outlined below.

ELIGIBILITY:
Inclusion criteria:

* Adult patients that are part of the regular healthcare patient flow at the investigational sites, or as separately invited to participate in this investigation.
* Patients with signed informed consent

Exclusion criteria:

* Cognitive impairment
* Patients unable to understand the oral and written study information in Swedish or English
* Other severe disorder or terminal disease, e.g. infection/sepsis, severe COPD or metastatic cancers.
* Patients unable to provide an informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study participants mainly consist of a prospective primary care population. All patients visiting the clinical sites, seeking care, or as separately invited, are offered to participate in this investigation. This includes sub-groups of patients with hypertension, valvular disease or risk for IHD.
  An extended investigation will be offered to participants judged to have an increased risk of cardiovascular disease in the primary care population, or for separately invited subjects with increased cardiovascular risk, known valvular disease, or as healthy controls. Repeated yearly measurements plan to be performed in interested subjects.
Sampling Method: Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between vibrometer-based PWV and ultrasound-based PWV | Typically same day or within 3-6 months of enrolment, at extended visit. If attending a 1-year follow-up, then around 1 year and 3-6 months from enrolment (follow-up extended visit).
  Vibrometer-based PWV in relation to ultrasound-based PWV, including both the carotid-femoral and aorto-femoral pathways. PWV in m/s, a measure of arterial stiffness.
Assess associations between vibrometer measurements and clinical measures of increased cardiovascular risk | Typically within 3 months of initial visit and enrolment, at extended visit. If attending a 1-year follow-up, then around 1 year and 3 months from enrolment.
  Vibrometer-derived PWV association with risk or presence of established atherosclerotic cardiovascular disease (ASCVD) based on ultrasound or clinical assessment.
Assess prediction performance of increased cardiovascular risk when combining vibrometer measurements, brachial BP, ABI and ECG in prediction models | Typically within 3-6 months of enrolment (extended visit). If attending a 1-year follow-up, then around 1 year and 3 months from enrolment (follow-up extended visit)..
  Combining vibrometer measurements, brachial BP, ABI, TBI and ECG in prediction models, may provide an improved prediction of increased cardiovascular risk (as defined above).
Assess performance of a multimodal risk score using data from the current study and the in parallel performed investigation "Spectrum 1" (CIV ID: CIV-22-07-039907). | Typically within 3-6 months after enrolment (extended visit). May include 1-year follow-up, in which case 1 year and 3-6 months (follow-up extended visit).
  Assess prediction of cardiovascular disease risk when adding parameters from the clinical study "Spectrum 1" to models based on parameters from the present study (vibrometer-based parameters, brachial BP, ABI, TBI, ECG).
  Outcome will be defined by presence of CVD risk or confirmed CVD based on ultrasound or clinical information, increased risk by risk scores, familial hypercholesterolemia, diabetes mellitus.
Assess associations between vibrometer measurements and presence of aortic valve pathology | Typically within 3-6 months of enrolment, at extended visit. If attending a 1-year follow-up, then around 1 year and 3-6 months from enrolment (follow-up extended visit).
  Vibrometer measurements, including left ventricular ejection time (LVET), in relation to aortic valve pathology, including aortic sclerosis, stenosis, or insufficiency, ranging from none to severe, and bicuspid aorta valve, assessed by ultrasound.
Assess associations between vibrometer measurements and ankle-brachial index | Typically at initial visit, same day as enrolment. If attending a 1-year follow-up, then around 1 year from enrolment.
  Vibrometer-derived PWV measurements in relation to increased risk for CVD as assessed by ankle-brachial index (ABI).
Assess associations between vibrometer measurements and measure of increased cardiovascular risk by risk score | Typically at initial visit, same day as enrolment. If attending a 1-year follow-up, then around 1 year from enrolment.
  Vibrometer-derived PWV measurements in relation to increased risk for CVD as assessed by established risk score (SCORE2).
  SCORE 2 is a risk prediction model to estimate 10-year risk of fatal or non-fatal atherosclerotic cardiovascular disease. Variables used in the model are age, sex, smoking status, systolic blood pressure and non-HDL cholesterol levels.

SECONDARY OUTCOMES:
Assess correlation between vibrometer-based PWV and other PWV reference methods | Typically same day as enrolment, or within 3-6 months of enrolment (extended visit). If 1-year follow-up, then within 1 year and 3-6 months from enrolment.
  Vibrometer-based PWV in relation to other reference methods for assessment of PWV, such as a single brachial-cuff based method (Arteriograph, Tensiomed), and peripheral piezo sensors (located on hands and feet). PWV in m/s, a measure of arterial stiffness.
Assess correlation between vibrometer-based LVET and ultrasound-based LVET | Typically same day or within 3-6 months of enrolment, at extended visit. If attending a 1-year follow-up, then around 1 year and 3-6 months from enrolment (follow-up extended visit).
  Vibrometer-based LVET as assessed by detection of systolic onset and end, in relation to ultrasound-based LVET as assessed by LVET measured directly at the left ventricular outflow tract.
Assess correlation between vibrometer-based LVET and aortic valve Vmax by ultrasound continuous doppler signal | Same day as enrolment, or within 3-6 months of enrolment (extended visit). If 1-year follow-up visit, then 1 year and 3-6 months from enrolment (follow-up extended visit).
  Vibrometer-based LVET as assessed by detection of systolic onset and end in relation to peak aortic jet velocity (Vmax) assessed by continuous doppler signal.
  Vmax is a measure of the speed at which blood travels across the aortic valve.
Association between prevalence of hypertension and cardiac output and peripheral resistance | Same day as enrolment, or typically within 3-6 months of enrolment, (extended visit). If attending a 1-year follow-up, then around 1 year and 3-6 months from enrolment (follow-up extended visit).
  Association between blood pressure and ultrasound-derived markers for cardiac output and peripheral resistance.
Assess associations between vibrometer measurements and measures of increased cardiovascular risk by pulse pressure | Typically at initial visit, same day as enrolment, or at extended visit. If attending a 1-year follow-up, then around 1 year from enrolment.
  Vibrometer-derived PWV measurements in relation to increased risk for CVD as assessed by pulse pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Hellqvist, MD, Principal Investigator — Neko Health AB
Locations (3):
- Sweden (3):
  - Atrium Health Care Centre, Stockholm
  - Neko Health Centre, Regeringsgatan, Stockholm
  - Neko Health Centre, Sibyllegatan, Stockholm

IPD SHARING:
Plan to Share IPD: No